CLINICAL TRIAL: NCT00402792
Title: A Randomized, Multicenter, Double-blind Study Comparing the Analgesic Efficacy and Safety of Extended-Release Hydrocodone/Acetaminophen (Vicodin CR®) to Placebo in Subjects With Acute Pain Following Bunionectomy
Brief Title: A Study of Extended-Release Hydrocodone/Acetaminophen (Vicodin CR®) in Subjects With Acute Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Andrea Best, DO, MPH, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M05-765
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Pain
Keywords: Acute pain following bunionectomy surgery
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: hydrocodone / acetaminophen extended release (Experimental)
  Interventions: Drug: Hydrocodone/Acetaminophen Extended-Release
- Arm 2: hydrocodone / acetaminophen extended release (Experimental)
  Interventions: Drug: Hydrocodone/Acetaminophen Extended Release
- Arm 3: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocodone/Acetaminophen Extended-Release — 1 tablet q 12 hours
  Other Names: ABT-712; hydrocodone / acetaminophen extended release
  Arms: Arm 1: hydrocodone / acetaminophen extended release
Drug: Hydrocodone/Acetaminophen Extended Release — 2 tablets q 12 hours
  Other Names: ABT-712; hydrocodone / acetaminophen extended release
  Arms: Arm 2: hydrocodone / acetaminophen extended release
Drug: Placebo — 2 tablets q 12 hours
  Arms: Arm 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness (level of pain control) and safety of the administration of Extended-Release Hydrocodone/Acetaminophen compared to placebo over a 48 hour dosing period in patients who have had bunionectomy surgery and to assess the safety of the drug for 7 days after patients are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 to 65
* Subject is scheduled to undergo primary, unilateral first metatarsal bunionectomy surgery
* Meet specific pain intensity criteria on the morning after surgery
* Willing to be confined for 4 days following surgery
* If female, must be of non-child bearing potential or practicing birth control

Exclusion Criteria:

* Is allergic to or has a serious reaction to hydrocodone, acetaminophen, lidocaine, propofol, morphine sulfate, oxycodone, and/or similar drugs
* Is allergic to or has a serious reaction to aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Has a history of certain gastrointestinal diseases that may narrow or slow down the gastrointestinal tract
* Has specific active or uncontrolled seizure disorders
* Has been diagnosed with certain cancers within the past 5 years
* Has a history of certain psychiatric disorders or requires treatment with certain drugs for depression
* Has specific clinically significant illnesses or laboratory abnormalities
* Has received corticosteroid treatment or any investigational drug within a specific timeframe

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Time-interval weighted sum of pain intensity difference (SPID) using the visual analog scale (VAS) for the 0 to 12 hour interval following study drug administration. | 12 hours
  Sum of pain intensity difference using a 100 mm Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Time-interval weighted sum of pain relief (TOTPAR) | 12 hours
Time-interval weighted sum of pain relief and pain intensity difference (SPRID) | 12 hours
Perceptible pain relief | 12 hours
Meaningful pain relief | 12 hours
Pain relief (PR) | 12 hours
Pain intensity (PI) | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, MD, Study Director — Abbott
Locations (5):
- United States (5):
  - Site Ref # / Investigator 2589, Austin, Texas
  - Site Ref # / Investigator 2587, Houston, Texas
  - Site Ref # / Investigator 2586, San Antonio, Texas
  - Site Ref # / Investigator 2588, San Marcos, Texas
  - Site Ref # / Investigator 2585, Salt Lake City, Utah